CLINICAL TRIAL: NCT00762749
Title: An Open-Label, Single-Dose Study Evaluating the Pharmacokinetics of Diphenhydramine in Children and Adolescents
Brief Title: Study to Evaluate Diphenhydramine in Children and Adolescents
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: DPHNCO1003
Record Dates: First submitted 2008-09-26; First posted 2008-09-30 (Estimated); Last update posted 2011-10-06 (Estimated); Status verified 2011-10

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic | interventions — Diphenhydramine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- diphenhydramine HCl (Experimental): diphenhydramine HCl / Children's Benadryl Allergy Liquid
  Interventions: Drug: diphenhydramine HCl

INTERVENTIONS:
Drug: diphenhydramine HCl — A single liquid dose of diphenhydramine HCl (12.5 mg /5 mL) followed by water, according to an age-weight dosing schedule
  Other Names: Children's Benadryl Allergy Liquid

SUMMARY:
To characterize the pharmacokinetics of diphenhydramine in two pediatric populations: children, ages 2 to < 12 years, and adolescents, ages 12 to < 18 years.

DETAILED DESCRIPTION:
This study has an open-label, single-dose classical pharmacokinetic design with no comparator treatment or group. Twenty-four (24) children, ages 2 to < 12 years, and 12 adolescents, ages 12 to < 18 years, with symptoms due to hay fever or other upper respiratory allergies will complete the study. To ensure that younger children are represented, at least 35% (8) of the children enrolled will range from 2 to < 6 years of age.

ELIGIBILITY:
Inclusion Criteria:

* Male and female children and adolescents, ages 2 to < 18 years, with a minimum weight of 24 pounds will be eligible to participate. In addition, each subject will be > 5th percentile and < 95th percentile for weight based on age and gender.
* Subjects will have a body mass index (BMI) > 5th percentile and less than or equal to 90th percentile for age and gender.
* Subjects who have a history of allergic rhinitis and who are experiencing symptoms due to hay fever or other upper respiratory allergies will be included.
* Subjects who do not use concurrent medications, except for low-dose inhaled glucocorticosteroids for allergic rhinitis or mild concurrent asthma, if dose is stabilized before entry in the study (ie, dose is not changed for 1 month prior to entry or during the study), and inhaled short-acting beta-2 adrenergic agonists for concomitant asthma, as needed;

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, or neurologic disease.
* Findings from the medical history or physical examination with vital sign measurements that are not within the range of clinical acceptability.
* Have a known sensitivity or allergy to diphenhydramine or EMLA cream.
* Have a known sensitivity or allergy to red dye.
* Have asthma symptoms at the time of study entry or requiring medications other than allowed in Inclusion Criterion 4;
* Took any prescription (other than allowed in Inclusion Criterion 4) or nonprescription medication, within seven days or five half-lives (whichever is longer) before the study's start date.
* Took any herbal supplements or drank grapefruit juice with 28 days of the study's start date.
* Participated in, or completed, another clinical trial within seven weeks before the study's start date.
* Have a history of drug, alcohol, and tobacco use (older children and adolescents)
* Have a history of hepatitis B, a previous positive test for hepatitis B surface antigen, or a previous positive hepatitis C antibody.
* Have a history of HIV infection or previous demonstration of HIV antibodies.
* Pregnant or nursing females; females of childbearing potential who are unwilling or unable to use an acceptable method of contraception from at least three months prior to the first dose of study medication until completion of follow-up procedures.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 36 (Actual)
Dates: Start 2008-09; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters | predose (0), and 0.5, 1, 1.5, 2, 4, 6, 8, 10, 12, and 24 hours after the dose

SECONDARY OUTCOMES:
Safety Assessments will consist of monitoring vital signs and all non-serious Adverse Events (AEs) and Serious Adverse Events (SAEs), their frequency, severity, seriousness, and relationship to the investigational product. | throughout duration of the study + 2 days (+ 30 days for spontaneously reported SAEs)

CONTACTS AND LOCATIONS:
Overall Officials: Cathy M Gelotte, PhD, Study Director — McNeil Consumer Healthcare Division of McNEIL-PPC, Inc.
Locations (1):
- Arkansas Medical Research Testing Center, Little Rock, Arkansas, United States